CLINICAL TRIAL: NCT04291833
Title: Prospective, Assessment of Vitamin D and Calcium Supplementation, Improvement of Nutritional Status and Preoperative Rehabilitation in Patients Before Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Bartlomiej Szpyra, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KBET/271/B/2014
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Knee Osteoarthritis; Vitamin D Deficiency; Pain, Postoperative; Arthropathy of Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Vitamin D Deficiency; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Active Comparator): Protein supplementation BID, Vitamin D and calcium supplementation Vitamin D 2000 IU / d, calcium 1000mg/d, exercise 6 months
  Interventions: Behavioral: Intervention group 1
- Intervention group 2 (Active Comparator): Protein supplementation QD, Vitamin D and calcium supplementation Vitamin D 1000 IU / d, calcium 500mg/d, exercise 3 months
  Interventions: Behavioral: Intervention group 2
- Control group 0 (Placebo Comparator): no protein supplementation , no Vitamin D and calcium supplementation , no exercise
  Interventions: Behavioral: Control group 0

INTERVENTIONS:
Behavioral: Intervention group 1 — Protein supplementation BID, Vitamin D and calcium supplementation Vitamin D 2000 IU / d, calcium 1000mg/d, exercise 6 months
  Arms: Intervention group 1
Behavioral: Intervention group 2 — Protein supplementation QD, Vitamin D and calcium supplementation Vitamin D 1000 IU / d, calcium 500mg/d, exercise 3 months
  Arms: Intervention group 2
Behavioral: Control group 0 — no protein supplementation , no Vitamin D and calcium supplementation , no exercise
  Arms: Control group 0

SUMMARY:
Prospective randomized study of 150 patients qualified for knee arthroplasty between 2015 and 2017. Patients were randomized into 3 groups receiving vitamin D and calcium supplementation, increased protein supply and preoperative rehabilitation, respectively.

Following factors were analyzed: changes in vitamin D3, calcium, total protein, albumin and CRP levels during preparation for surgery, nutritional status on the Subjective Global Assessment (SGA) scale, osteoporosis risk assessment according to the Osteoporosis Risk SCORE, level of pain felt on the scale VAS and the number of analgesics used, the result of the Duke Activity Status Index, the result of the following scales: Cardiac Risk Index for Orthopedic Surgery (Lee), Knee injury and Osteoarthritis Outcome Score (KOOS), Fear Avoidance Beliefs Questionnaire (FABQ) about Physical Activity, The Quality of Life Scale (QOLS). Additionally, the occurrence of perioperative complications was analyzed (e.g. venous thrombosis and pulmonary embolism, wound or joint infection, excessive bleeding, loosening of the implant, bone fracture or fracture, pain).

ELIGIBILITY:
Inclusion Criteria:

* with a disease lasting more than 5 years and without total limitation of physical fitness,
* reporting pain> 5 on the VAS scale (Visual Analogue Scale)
* general fitness according to the ASA (Amercican Society of Anestesiology) scale up to 3

Exclusion Criteria:

* patients with metabolic and systemic disorders with contraindications for calcium substitution, vitamin D3 and protein supply,
* intolerance of physical effort> 2, 5 MET (Metabolic Equivalent of Task)
* limitation of the degree overall efficiency> 3 in the ASA classification

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Pain control satisfaction assessed on the Visual Analogue Scale (VAS) | 18 months
  Visual Analogue Scale (VAS) is a measure determining the intensity of pain by means of a visual analogue scale. Subject is marking the examined point on a line of 10 cm long, where the value 0 is assigned the total absence of pain, and 10 the strongest pain that can be imagined.
Vitamin D concentration in blood, based on laboratory analysis. | 18 months
  Concentration of vitamin D in blood is a laboratory parameter, measured in unit of ng/ml. Levels below 20 ng/ml is a severe vitamin D deficiency condition that requires treatment. The result in the range 20-30 ng/ml means that the vitamin level is not sufficient. Values between 30-50 ng/ml are considered normal. This is one of the basic laboratory parameters for assessing the body's bone mineral metabilism.
Efficiency of the knee joint assessed on The Knee Injury and Osteoarthritis Outcome Score (KOOS) scale. | 18 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.

SECONDARY OUTCOMES:
Calcium ionized concentration in blood, based on laboratory analysis. | 18 months
  Calcium ionized concentration in blood is a laboratory parameter, measured in unit of mmol/l. The results below 1.16 mmol/l mean that the level is not sufficient, condition called hypocalcemia. Values between 1.16-1.32 mmol/l are considered normal. The results above 1.32 mmol/l mean hypercalcemia occurs. This is one of the basic laboratory parameters for assessing the body's bone mineral metabilism.
Total protein concentration in blood, based on laboratory analysis. | 18 months
  Total protein concentration in blood is a laboratory parameter, measured in unit of g/l. The results below 60 g/l mean that the level is not sufficient, condition called hypoproteinemia. Values between 60-80 g/l are considered normal. The results above 80 g/l mean hyperproteinemia occurs. This is one of the basic laboratory parameters for assessing the body's nutritional status.
Albumin concentration in blood, based on laboratory analysis | 18 months
  Albumin concentration in blood is a laboratory parameter, measured in unit of mg/ml. The results below 35 mg/l mean that the level is not sufficient, condition called hypoalbuminemia. Values between 35-50 mg/ml are considered normal. The results above 50mg/l mean hyperalbuminemia occurs. This is one of the basic laboratory parameters for assessing the body's nutritional status.
C-reactive protein (CRP) concentration in blood, based on laboratory analysis | 18 months
  C-reactive protein concentration in blood is a laboratory parameter, measured in unit of mg/l. The results below 5 mg/l are considered normal. The results above 5mg/l mean infection, trauma, stress or other aggravating factor. This is the major laboratory parameter for assessing homeostatic balance.
Efficacy of protein supplementation assessed on the Subjective Global Assessment (SGA) scale. | 18 months
  Subjective global assessment (SGA) is the gold standard for diagnosing malnutrition. SGA is a simple bedside questionnaire method used to diagnose malnutrition and identify those who would benefit from nutrition care. The assessment includes taking a history of recent intake, weight change, gastrointestinal symptoms and a clinical evaluation. Results are on a scale from 1 to 7. Values 1 and 2 means high risk of malnutririon, from 3 do 5 medium risk, and from 6 do 7 mild risk.
Efficacy of vitamin D and calcium supplementation assessed on the Simple Calculated Osteoporosis Risk Estimation (SCORE) scale. | 18 months
  Simple Calculated Osteoporosis Risk Estimation (SCORE) scale is the questionnaire tool for diagnosing Osteoporosis risk. It has been reported to appropriately identify person who should be referred for bone densitometry. Results are on a scale from 0 to 50 points. Points from 16 to 50 means high risk of osteoporosis , points from 7 to 15 moderate risk and from 0 do 6 low risk of osteoporosis.
Acceptability of physical activity based on Duke Activity Status Index (DASI) scale. | 18 months
  The Duke Activity Status Index is a self-administered questionnaire that measures a patient's functional capacity. It can be used to get a rough estimate of a patient's peak oxygen uptake. Results are on a scale from 0 to 57,95 points. The higher the score, the more intense the acceptable physical activity.
Incidence of cardiovascular hazard based on Cardiac Risk Index for Orthopedic Surgery (Lee) scale. | 18 months
  Cardiac Risk Index for Orthopedic Surgery (Lee) is the questionnaire tool for diagnosing cardiovascular hazard in orthopedics patients. Results are on a scale from 0 to 6 points. Points from 3 to 6 means estimated risk of 4%, 2 points is 2,3% of risk, 1 point is 1,7% of risk and 0 points means less than 1 % of cardiovascular event.
Unwillingness of phisical activity due to pain based on Fear Avoidance Beliefs Questionnaire (FABQ) scale. | 18 months
  Fear Avoidance Beliefs Questionnaire (FABQ) scale is a questionnaire based on the Fear-Avoidance Model of Exaggerated Pain Perception, a model created in attempts to explain why some patients with acute painful conditions can recover while other patients develop chronic pain from such conditions. The FABQ focuses specifically on how a patient's fear-avoidance beliefs about physical activity and work. It consists of 16 questions scaled form 0 do 6, higher score indicates fear avoidance behaviors.
The Quality of Life based on The Quality of Life (QOLS) scale. | 18 months
  The Quality of Life (QOLS) scale is the most known scale measures factors like satisfaction, perceptions of control, involvement, commitment, and work-life balance, in terms of one's personal perception. QOLS has 16 items, scaled form 1 do 7, higher score indicates superior appraisal of each aspect of life.
Incidence of Treatment-Emergent Adverse Events (AE) as assessed by frequency. | 18 months
  Incidence of Adverse Events (AE) was summed up and analyzed in each group. They were divided into 7 groups.
  1. - a serous wound leak requiring albumin transfusion
  2. - bleeding that requires RBC transfusion
  3. - perioperative infection
  4. - postoperative infection
  5. - pulmonary embolism
  6. - other
  7. - death. Every case was appropriately assigned, analyzed and evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartlomiej Szpyra, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: No